CLINICAL TRIAL: NCT06873789
Title: A Phase 1/2, Open-Label, Multicenter Study of INCB177054 in Participants With Select Advanced or Metastatic Solid Tumors
Brief Title: A Study to Evaluate INCB177054 in Participants With Select Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB177054-101
Record Dates: First submitted 2025-03-11; First posted 2025-03-13 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors; Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Solid Tumors; INCB177054

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1a: Dose Escalation monotherapy (Experimental): INCB177054 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB177054
- Part 1b: Pharmacodynamic cohort (Experimental): INCB177054 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB177054
- Part 1c: Dose Expansion monotherapy (Experimental): INCB177054 at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB177054
- Part 2a: Dose Escalation combination (Experimental): INCB177054 in combination with retifanlimab at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB177054; Drug: Retifanlimab
- Part 2b: Dose Expansion combination (Experimental): INCB177054 in combination with retifanlimab at the protocol-defined dose strength based on cohort assignment.
  Interventions: Drug: INCB177054; Drug: Retifanlimab

INTERVENTIONS:
Drug: INCB177054 — INCB177054 will be administered at protocol defined dose.
Drug: Retifanlimab — Retifanlimab will be administered at protocol defined dose.
  Arms: Part 2a: Dose Escalation combination; Part 2b: Dose Expansion combination

SUMMARY:
This study will be conducted to evaluate INCB177054 given as monotherapy or in combination with retifanlimab in participants with select advanced or metastatic solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated life expectancy greater than 12 weeks.
* ECOG performance status score of 0 or 1.
* Measurable disease per RECIST v1.1 on CT or MRI.
* Part 1a and 2a (dose escalation) and Part 1c (dose expansion): participants who have a confirmed tissue diagnosis of a solid malignant tumor that is progressing and not amenable to curative surgery or other curative treatment modalities.

  * Part 1a (monotherapy): Participants must have had disease progression on/after prior treatment and have been considered for all standard available therapies (have disease progression on all available standard treatment options or are intolerant or ineligible to them or has refused available options approved in the region).
  * Part 2a (combination): participants with advanced malignant tumors for whom immunotherapy is an appropriate treatment option.
* Part 1b incurable locally recurrent or metastatic HNSCC:

  * Tissue diagnosis of HNSCC.
  * Locally recurrent disease must not be amenable to therapy (surgery and/or radiation therapy with or without chemotherapy) with curative intent. Participants who refuse curative salvage surgery for locally recurrent disease are ineligible.
  * Eligible primary tumor locations include oral cavity, oropharynx, hypopharynx, or larynx. Primary tumors of the nasopharynx, sinonasal cavity, or salivary gland are excluded.
* Part 2b combination dose-expansion cohorts in locally advanced or metastatic SCAC (Group 1), metastatic PD-L1-positive (TPS ≥ 50%) NSCLC (Group 2), or locally recurrent or metastatic PD-L1-positive (CPS ≥ 1%) HNSCC (Group 3) (Primary tumors of the nasopharynx, sinonasal cavity, or salivary gland are excluded).
* Availability of a baseline archival tumor specimen or willingness to undergo a pretreatment biopsy to obtain.
* If HIV-positive, CD4+ count must be greater than or equal to 350 cells/μL, must have undetectable viral load per standard of care assay, and receiving antiretroviral therapy not containing a moderate or potent CYP3A4/CYP3A5 inhibitor or inducer for at least 4 weeks prior to study enrollment, and have not had any HIV-related opportunistic infection for at least 4 weeks prior to study enrollment.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Known additional invasive malignancy within 1 year of the first dose of study drug.
* Known active CNS metastases and/or carcinomatous meningitis and/or leptomeningeal disease, or evidence of progression of previously treated CNS metastases.
* Prior treatment with a DGK inhibitor.
* Receipt of anticancer medications, investigational drugs, or other interventional clinical studies within 5 half-lives or 28 days before the first administration of study drug.
* History of organ transplant, including allogeneic stem cell transplantation.
* Radiation therapy administered within 28 days of the start of treatment.
* Any residual toxic effects ≥ Grade 2 from prior therapy or surgery.
* Any immune-related toxicity during prior immune therapy for which permanent discontinuation or prolonged immunosuppression was recommended to manage.
* Laboratory values specified at screening.
* Significant concurrent, uncontrolled medical conditions, including but not limited to hepatic, gastrointestinal conditions, pulmonary, cardiovascular, and active autoimmune disease.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment.
* Active HBV or HCV.
* Prohibited medication per protocol.
* Hypersensitivity to any component of study treatment or formulation components.
* Women who are pregnant or breastfeeding.
* Has received a live vaccine within 28 days of the planned start of study treatment.
* Any condition that would interfere with participation.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 12 months and 45 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Number of participants with TEAEs leading to study drug modifications | Up to approximately 12 months and 45 days
  Number of participants with TEAEs leading to dose modification including interruptions, dose reductions, and discontinuation of study drug.

SECONDARY OUTCOMES:
Objective Response | Up to approximately 12 months
  Defined as having a best overall response of Complete Response (CR) or Partial Response (PR) by investigator assessment (all participants) per RECIST v1.1.
Duration of Response | Up to approximately 12 months
  Defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression as determined by the investigator by radiographic disease assessment per RECIST v1.1 or death due to any cause if occurring sooner than progression.
Disease Control | Up to approximately 12 months
  Defined as having a best overall response of CR, PR, or Stable Disease (SD), by investigator assessment per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (9):
- United States (9):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Valkyrie Clinical Trials, Panorama City, California
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Cancer and Hematology Centers of Western Michigan-Start Midwest, Grand Rapids, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Carolina Bio Oncology, Huntersville, North Carolina
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Upmc Cancercenter, Pittsburgh, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A study to evaluate INCB177054 in Participants With Select Advanced or Metastatic Solid Tumors — https://www.incyteclinicaltrials.com/study/?id=INCB177054-101&SearchTerm=INCB177054-101&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=